CLINICAL TRIAL: NCT07202104
Title: Improvement of an Algorithm to Detect Structural Heart Murmurs in Adult Patients Using Electronic Stethoscopes
Status: Recruiting | Type: Observational
Sponsor: Eko Devices, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025.1
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Structural Heart Disease
Keywords: structural heart disease; structural murmur

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Eko digital stethoscopes — Use of the Eko CORE 500 digital stethoscope and 3M Littmann CORE Digital Stethoscope to auscultate and record cardiac phonocardiogram and (when available) electrocardiogram waveforms, as well as heart sounds.

SUMMARY:
The main objective of this study is to evaluate a machine learning model's ability to detect murmurs indicative of structural heart disease ("structural murmur") by analyzing phonocardiogram waveforms-and simultaneous electrocardiogram waveforms when available-in multiple auscultatory positions per subject. Diagnosis of structural murmur will be confirmed by gold-standard echocardiography and reviewed by an expert panel of cardiologists.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Patient or patient's legal healthcare proxy consents to participation
* Documented history of SHD
* Undergoing (or has undergone, within 30 days) a complete echocardiogram
* Willing to have heart recordings done with two different electronic stethoscopes

Exclusion Criteria:

* Patient or proxy is unwilling/unable to give written informed consent
* Unable to complete a complete echocardiogram, or none recent completed within the last 30 days
* No documented history of SHD
* Experiencing a known or suspected acute cardiac event
* Mechanical ventricular support (such as ECMO, LVAD, RVAD, BiVAD, Impella, intra-aortic balloon pumps, TAH, VentrAssist, DuraHeart, HVAD, EVAHEART LVAS, HeartMate, Jarvik 2000)
* Unwilling or unable to follow or complete study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be screened for eligibility from cardiology clinics, echocardiogram clinics, and inpatient areas. In order to be eligible, a patient must be 18+ years of age, have a documented history of structural heart disease, and has undergone an echocardiogram within the last 30 days. If a patient meets all of the specified inclusion criteria, and none of the specified exclusion criteria, the patient or their proxy will be approached to discuss participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 6 months
  Evaluate a machine learning model's ability to detect murmurs indicative of structural heart disease ("structural murmur") by analyzing phonocardiogram waveforms-and simultaneous electrocardiogram waveforms when available-in multiple auscultatory positions per subject. Diagnosis of structural murmur will be confirmed by gold-standard echocardiography and review by an expert panel of cardiologists.

CONTACTS AND LOCATIONS:
Locations (1):
- Cox Medical Centers, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No